CLINICAL TRIAL: NCT03414814
Title: Phase II Study of Osimertinib in NSCLC Patients With EGFR Exon 20 Insertion Mutation
Brief Title: Osimertinib for NSCLC With EGFR Exon 20 Insertion Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: AstraZeneca (Industry); Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Tae Min Kim, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG LU17-19
Record Dates: First submitted 2017-12-21; First posted 2018-01-30 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced or Metastatic NSCLC
Keywords: NSCLC; Osimertinib; EGFR exon 20 insertion mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Osimertinib (Experimental): Osimertinib at 80mg dose will be administered orally once daily.
  Interventions: Drug: Osimertinib 80 MG [Tagrisso]

INTERVENTIONS:
Drug: Osimertinib 80 MG [Tagrisso] — Osimertinib 80mg once daily until disease progression

SUMMARY:
This is a single-arm, non-randomized multicentre phase 2 study in NSCLC patients with EGFR exon 20 insertion mutation, whose disease has progressed on standard chemotherapy.

DETAILED DESCRIPTION:
EGFR exon 20 insertion-mutant NSCLCs are generally resistant to 1st-generation EGFR tyrosine kinase inhibitors (TKIs) as well as 2nd-generation EGFR TKIs (overall response rates of 0-8.7%). Osimertinib is an oral, potent, irreversible EGFR-TKI selective for sensitizing EGFR and EGFR T790M resistance mutations with a significant selectivity margin against wild-type EGFR. Osimertinib is potent with a wide therapeutic window in Ba/F3 cells with EGFR exon 20 insertion mutations. Therefore, this study will be performed to investigate the efficacy of osimertinib in NSCLC patients with EGFR exon 20 insertion mutation

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male or female must be > 19 years of age.
3. Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy with local confirmation of the presence of the EGFR exon 20 insertion mutation
4. Disease progression while on standard chemotherapy (platinum doublet chemotherapy or single-agent chemotherapy in selected patients)
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Patients must have a life expectancy ≥ 12 weeks
7. Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:
8. Male patients should be willing to use barrier contraception
9. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
10. At least one measurable lesion
11. Provision of archival FFPE tissue
12. Provision of informed consent for translational genetic research

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both sponsor staff and/or staff at the study site)
2. Previous treatment with osimertinib (3rd generation EGFR TKIs such as olumtinib, EGF816 etc)
3. Treatment with an investigational drug within five half-lives of the compound
4. Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inhibitors of CYP3A4 (at least 1 week prior) and potent inducers of CYP3A4 (at least 3 week prior) (Appendix A). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer/inhibitory effects on CYP3A4.
5. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy.
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
7. Patients with symptomatic CNS metastases who are neurologically unstable; however, those with asymptomatic CNS metastases who do not require steroids for at least 4 weeks prior to start of osimertinib are eligible.
8. Past medical history of ILD, drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
9. Inadequate bone marrow reserve or organ function
10. QTc prolongation (mean resting corrected QTc > 470 msec)
11. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib
12. History of hypersensitivity to osimertinib (or drugs with a similar chemical structure or class to osimertinib) or any excipients of these agents
13. Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry
14. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
15. Previous allogeneic bone marrow transplant.
16. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae Min Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim YJ, Kim S, Kim TM, Suh KJ, Kim M, Kim SH, Keam B, Kim DW, Lee JS, Heo DS. A phase II study of osimertinib in patients with NSCLC harboring EGFR exon 20 insertion: A multicenter trial of the Korean Cancer Study Group (LU17-19). Lung Cancer. 2024 Aug;194:107870. doi: 10.1016/j.lungcan.2024.107870. Epub 2024 Jul 3. PMID 38986212

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Osimertinib
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with NSCLC harboring EGFR exon 20 insertions
Arm/Group | Osimertinib
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 61 [42 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 15

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Investigator-assessed, confirmed objective response by RECIST version 1.1
Time Frame: Until study completion, from date of initiation until the date of first documented progression, unacceptable toxicities or withdrawl, whichever came first. (upto about 29months)
Population: The proportion of patients who had complete reponse (CR) and partial reponse (PR) as the best response among 80mg osimertinib administered 15 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 15
Participants | 0

2. Secondary Outcome: Serious Adverse Events
Description: AEs/SAEs as defined by NCI CTCAE version 4.0
Time Frame: From date of initiation until the date of first documented progression, unacceptable toxicities or withdrawal, whichever came first. Until study completion. (upto about 29months)
Measure: Number; unit: cases
Arm/Group | Osimertinib
Number analyzed (Participants) | 15
cases
  General weakness | 1
  Acute urinary retention | 1
  Pneumonia | 2
  Colitis | 1
  Azotemia | 1
  Hypercalcemia | 1
  Femur fracture | 1

3. Secondary Outcome: Progression-free Survival
Description: PFS as defined by RECIST version 1.1
Time Frame: From date of initiation until the date of first documented progression, unacceptable toxicities or withdrawl, whichever came first. Until study completion. (upto about 29months)
Population: The PFS rate at the time of data cutoff (10 June 2020) for 80mg osimertinib administered 15 patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Osimertinib
Number analyzed (Participants) | 15
months | 3.8 [1.7 to 5.5]

4. Secondary Outcome: Overall Survival
Description: OS as defined by RECIST version 1.1. The time from the first date of IP administration to the date of death.
Time Frame: From the first date of IP administration to the date of death. (upto about 29months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Osimertinib
Number analyzed (Participants) | 15
months | 6.5 [3.9 to 29]

ADVERSE EVENTS:
Time Frame: from the day of first IP administration to 30 days after the last IP administration (till PD or unacceptable toxicity), (upto about 29months)
Arm/Group | Osimertinib
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 8/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osimertinib (N=15)
Colitis (Gastrointestinal disorders) | 1 (1)
Azotemia (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
General weakness (General disorders) | 1 (1)
Acute urinary retention (Renal and urinary disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osimertinib (N=15)
Dry eye (Eye disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Asthenia (General disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Localised oedema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT03414814/Prot_SAP_000.pdf